CLINICAL TRIAL: NCT04973436
Title: Dialectical Behavioral Therapy Skills Training for Metastatic Lung Cancer Patients
Brief Title: DBT for Metastatic Lung Cancer
Acronym: LiveWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108640
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer Metastatic
Keywords: dialectical behavioral therapy skills training; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol (Experimental): The intervention, "LiveWell" will teach participants dialectical behavioral therapy-based skills to reduce psychological distress through improved physical symptom management, emotion regulation, and tolerance of uncertainty. Informed by feedback from patients and providers collected in Phase of of the study, the LiveWell intervention consists of of 8 sessions delivered one-on-one, approximately weekly. Sessions will last approximately 45-60 minutes each.
  Interventions: Behavioral: Dialectical Behavioral Therapy Skills Training

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy Skills Training — LiveWell: Dialectical behavioral therapy skills training adapted for patients with metastatic lung cancer

SUMMARY:
Metastatic lung cancer patients experience significantly greater psychological distress (i.e., depression, anxiety) compared to other cancers. Psychological distress is as a prognostic indicator for worse clinical outcomes and poorer overall survival in cancer patients. Dialectical behavioral therapy (DBT) is a trans-diagnostic, evidence-based psychotherapy that teaches participants a core set of behavioral skills (distress tolerance, emotion regulation, mindfulness, interpersonal effectiveness) to cope more effectively with emotional and physical symptoms. The proposed study seeks to adapt and pilot test DBT skills training for patients with metastatic lung cancer using the ADAPT-ITT framework. Participants will be metastatic lung cancer patients who score >=3 on the National Comprehensive Cancer Network distress thermometer. Phase I aims to use focus groups and interviews with key stakeholders (metastatic lung cancer patients (N=20), thoracic oncology providers (N=6), clinicians with expertise in survivorship and behavioral symptom management (N=6)) to determine if and how DBT skills training must be modified for implementation with metastatic lung cancer patients. Adapted material will be reviewed by topical experts in DBT and implementation science to produce a manualized, adapted DBT skills training protocol for metastatic lung cancer patients (LiveWell). Phase II aims to pilot test LiveWell (N=30) to assess feasibility, acceptability, and examine pre-to-post intervention outcomes of psychological distress, (i.e., depression and anxiety) fatigue, dyspnea, pain, emotion regulation, tolerance of uncertainty, and DBT coping skill use. LiveWell will consist of coping skills training sessions delivered either in-person or via videoconferencing technology. Study measures will be collected at baseline, immediately post-intervention, and 1-month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. be diagnosed with metastatic (AJCC stage IV) non-small cell lung cancer
2. be undergoing systemic treatment (chemotherapy, targeted therapy, and/or immunotherapy) for lung cancer at Duke Cancer Institute
3. score >3 on the National Comprehensive Cancer Network Distress Thermometer for distress over the past week (Range: 0-10)
4. be > 18 years of age
5. be able to understand, speak, and read English
6. be able to provide informed consent

Exclusion Criteria:

1. reported or suspected cognitive impairment subsequently informed by a Montreal Cognitive Assessment (MOCA) of <26
2. presence of untreated serious mental illness (e.g., schizophrenia) indicated by the medical chart, treating oncologist, or other medical provider
3. expected survival of 4 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Somers, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hyland KA, Neacsiu AD, Fisher HM, Cowperthwait CM, Chou N, Stinchcombe TE, Oeffinger KC, Porter LS, Dorfman CS, Keefe FJ, Somers TJ. LiveWell: Pilot Feasibility Trial of an Adapted Dialectical Behavioral Therapy Skills Training Protocol in Patients With Metastatic Non-Small Cell Lung Cancer. Psychooncology. 2025 Dec;34(12):e70357. doi: 10.1002/pon.70357. PMID 41392376

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was lost to contact prior to baseline assessment.
Period: Overall Study
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Started | 30
Completed Protocol | 27
Post-Intervention Assessment | 26
1-Month Follow-up Assessment | 24
Completed | 24
Not Completed | 6
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Time since lung cancer diagnosis [Mean (Standard Deviation); unit: years] | 4.62 (4.06)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Study Accrual
Description: Treatment feasibility will be shown by meeting study accrual target (N = 30 for single-arm pilot)
Time Frame: Post-intervention (approximately 8 weeks)
Population: Individuals who were eligible for consent.
Measure: Count of Participants; unit: Participants
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 34
Participants | 31

2. Primary Outcome: Adherence as Measured by Number of Participants Who Completed All Intervention Sessions
Description: Adherence will be shown by at least 80% of intervention sessions completed.
Time Frame: Post-intervention (approximately 8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
Participants | 27

3. Primary Outcome: Feasibility as Measured by Number of Participants Lost From the Study Over Time
Description: Treatment feasibility will be shown by no more than 25% study attrition.
Time Frame: Post-intervention (approximately 8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
Participants | 4

4. Primary Outcome: Acceptability as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: CSQ items are rated on a 4-point scale from 1 (quite dissatisfied) to 4 (very satisfied), then averaged to obtain an overall acceptability score. Acceptability was demonstrated by >80% of participants reporting intervention satisfaction (an average CSQ score of 3 to 4). Reported as the number of participants who had an average CSQ score of 3 to 4.
Time Frame: Post-intervention (approximately 8 weeks)
Population: Participants who completed the CSQ.
Measure: Count of Participants; unit: Participants
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 26
Participants | 25

5. Primary Outcome: Psychological Distress as Measured by the PROMIS Depression Short Form Scales
Description: Distress will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (8 items) Short Form Scale. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater distress.
Time Frame: Baseline, post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the PROMIS Depression Short Form Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 51.82 (9.16)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 48.85 (8.69)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 48.18 (9.73)

6. Primary Outcome: Psychological Distress as Measured by the PROMIS Anxiety Short Form Scales
Description: Distress will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety (7 items) Short Form Scale. PROMIS scores are expressed as T-scores, with a mean of 50 and a standard deviation of 10. Higher scores indicate greater distress.
Time Frame: Baseline, post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the PROMIS Anxiety Short Form Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 29
score on a scale
  Baseline | 54.03 (8.25)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 51.75 (7.51)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 48.39 (8.82)

7. Secondary Outcome: Fatigue Severity as Measured by the Fatigue Symptom Inventory (FSI)
Description: Fatigue (i.e., severity and interference) will be assessed using the Fatigue Symptom Inventory (FSI). The FSI has a score range of 0 to 10, where a higher score indicates more fatigue.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the FSI.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 3.86 (1.80)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 3.36 (2.03)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 3.14 (2.24)

8. Secondary Outcome: Change in Dyspnea
Description: Breathlessness will be assessed using the Modified Medical Research Council Dyspnea Scale (MMRCDS). The MMRCDS has a score range of 0 to 4, where a higher score indicates worse dyspnea.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the MMRCDS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 0.97 (0.87)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 1.20 (1.08)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 1.00 (1.02)

9. Secondary Outcome: Pain Severity as Measured by the Brief Pain Inventory-Short Form (BPI-SF)
Description: The BPI-SF has a score range of 0 to 10, where a higher score indicates greater pain severity.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the BPI-SF.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 1.84 (1.80)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 1.48 (1.78)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 1.74 (1.97)

10. Secondary Outcome: Pain Interference as Measured by the Brief Pain Inventory-Short Form (BPI-SF)
Description: The BPI-SF has a score range of 0 to 10, where a higher score indicates greater pain interference.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the BPI-SF.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 1.99 (2.06)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 1.91 (2.36)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 1.64 (2.01)

11. Secondary Outcome: Change in Emotion Regulation as Measured by the Emotion Regulation Scale (DERS-18)
Description: The Difficulties in Emotion Regulation Scale (DERS-18) will be used to assess emotion regulation. The DERS-18 has a score range of 18-80, where a higher score indicates greater difficulty with regulating emotions.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 18, week 12)
Population: Participants who completed the DERS-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 32.33 (9.75)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 28.73 (7.57)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 27.96 (7.50)

12. Secondary Outcome: Change in Intolerance of Uncertainty as Measured by the Intolerance of Uncertainty Short Form (IUS)
Description: The Intolerance of Uncertainty Short Form (IUS) will be used to measure emotional, cognitive, and behavioral reactions to uncertain situations. The IUS has a score range of 12-60, where a higher score indicates greater intolerance of uncertainty.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the IUS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 25.50 (7.89)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 20.62 (4.82)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 20.88 (7.12)

13. Secondary Outcome: Change in Dialectical Behavioral Therapy (DBT) Skill Use as Measured by the DBT Ways of Coping Checklist (DBT-WCCL) -DBT Skills Subscale (DSS)
Description: The DBT Ways of Coping Checklist (DBT-WCCL) -DBT Skills Subscale (DSS) will be used to assess patient-reported frequency of skill use to manage difficult situations. The DBT-WCCL has a score range of 0 to 4, where a higher score indicates greater DBT skill use.
Time Frame: Baseline, post-intervention, one month post-intervention (approximately week 0, week 8, week 12)
Population: Participants who completed the DBT-WCCL-DSS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
Number analyzed (Participants) | 30
score on a scale
  Baseline | 1.95 (0.44)
  Week 8: number analyzed (Participants) | 26
  Week 8 | 2.24 (0.44)
  Week 12: number analyzed (Participants) | 24
  Week 12 | 2.25 (0.43)

ADVERSE EVENTS:
Time Frame: Up to approximately 16 weeks
Arm/Group | LiveWell: A Dialectical Behavioral Therapy Skills Training Protocol
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04973436/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04973436/ICF_000.pdf